CLINICAL TRIAL: NCT06252909
Title: Treating Common Mental Disorders in Women in Mozambique by Addressing Intimate Partner Violence in Couples
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Jennifer Mootz, Assistant Professor of Clinical Medical Psychology (in Psychiatry), New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23MH122661 (NIH)
Record Dates: First submitted 2024-01-24; First posted 2024-02-12 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-05

CONDITIONS: Depression; Anxiety; PTSD; Intimate Partner Violence
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Interpersonal Psychotherapy; Family Characteristics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interpersonal Psychotherapy for Couples (Experimental)
  Interventions: Behavioral: Interpersonal Psychotherapy for Couples
- Interpersonal Psychotherapy (Individual) (Active Comparator)
  Interventions: Behavioral: Interpersonal Psychotherapy (Individual)

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy for Couples — Interpersonal Psychotherapy for Couples (IPT-C) consists of 8 weekly conjoint sessions. The clinical goals are to "promote resolution of the role dispute via renegotiation of role relations between the marriage partners" and improve common mental disorders in the woman. Like Interpersonal Psychotherapy, IPT-C has an initiation phase (Session 1-2), middle phase (Sessions 3-6), and termination phase (Sessions 7-8).
  Arms: Interpersonal Psychotherapy for Couples
Behavioral: Interpersonal Psychotherapy (Individual) — Interpersonal Psychotherapy (IPT) is an evidence-based treatment to reduce depression and other common mental disorders. It focuses on helping patients resolve interpersonal problems of disagreements, loneliness, life changes, and grief, and/or change their orientation to the problem.
  Arms: Interpersonal Psychotherapy (Individual)

SUMMARY:
Adapting mental health treatments to address modifiable interpersonal problems has the potential to improve and sustain outcomes in low-resource settings where treatment gaps persist. This K23 Award will prepare the candidate to become an independent investigator with high-impact public health research and expertise in couple-based interventions that address interrelated mental health problems and intimate partner violence in couples by gaining expertise in engagement and treatment of men, adapting an evidence-based treatment for common mental disorders to address IPV in couples, designing and conducting randomized controlled trials with couples, and professional skills development. This work has applicability for low-resource low-income countries and US populations that experience couple-based violence and the mental health treatment gap. With its focus on intimate partners, the intervention also has the potential to benefit health and wellbeing of children.

ELIGIBILITY:
Inclusion Criteria:

* Both partners aged ≥18;
* both partners identify each other as one of (in case of polygamous marriage) their primary sexual partners of the opposite sex;
* partnered for at least 3 months;
* woman screens positive for a CMD using the Mental Wellness Tool developed and validated by our PRIDE team in Mozambique;
* couples have mild to moderate forms of situational IPV (Ongoing Abuse Scale score = 1 or above). See below exclusion criteria for how severity will be determined.;
* both partners desire to maintain the relationship;
* woman identifies marital dispute as the main interpersonal problem area causing CMD symptoms.

Exclusion Criteria:

* Any indicators of severe IPV. The determination of severity will be assessed using items (presence or absence) on the Conflict Tactics Scale (CTS). If any couple member answers yes to both of the following items: "I punched or hit my partner with something that could hurt" and "I kicked my partner," couples will be excluded. Couple members who answer yes to any of the following items: "I used a knife or gun on my partner," "I choked my partner," "I slammed my partner against a wall," "I beat up my partner," "I burned or scalded my partner on purpose," will be excluded. Finally, if any couple member reports that a violent behavior was repeated at least six times in a year by their partner or themselves, violence will be considered severe.;
* (2) discrepancy (>2) in reporting of frequency of violence on CTS in overall average scores of the partners or for any single behavior in the scale. For example, if the female partner reports that her male partner slapped her three times, but the male partner reports that he never slapped his female partner, the couple will be excluded for discrepant reporting for the act of slapping.;
* history of violent legal offences;
* male partner has severe CMD symptoms (PHQ-9 score of 20 or above; GAD-7 score of 15 or above; and PCL-C score of 45 or above); and either partner demonstrates/reports
* serious mental illness,
* cognitive impairment,
* history of mania (Psychosis Screening Questionnaire score = 1),
* hazardous alcohol use (AUDIT score of 8 or above),
* current suicidality,
* not speaking Portuguese,
* feeling unsafe to participate,
* inability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible women and their male partners will be recruited for this study.
Enrollment: 108 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire Client Satisfaction Questionnaire - 8 (CSQ-8) | measured at week 8
  The Client Satisfaction Questionnaire - 8 measures respondents' opinions about services they have received. Responses are based on a four-point scale (ranging from very negative to very positive), but the options differ depending on the item. Scores range from 8 to 32; higher values indicate higher satisfaction. Scores are calculated by summing scores across all items.
IPT Fidelity Checklist | measured up to 8 weeks
  The IPT Fidelity Checklist measures provider fidelity to Interpersonal Therapy. Providers are assessed for low (1), moderate (2), or high (3) adherence to each treatment element. A total score is calculated y summing individuals items. The PRIDE team has adapted this Checklist for Interpersonal Counseling, which will be further adapted in the proposed study for couple-based treatment.
Mental Wellness Tool | measured at pre-treatment and weeks 8, 12, 20, 32
  The Mental Wellness Tool was developed and validated by the PRIDE team in Mozambique to screen for and differentiate cases according to presence or absence of common mental disorders, severe mental illness, substance use disorders, and suicidal risk. Patients are asked three initial questions. If they respond positively to any of the 3 items, they are asked 10 additional items. The Mental Wellness Tool will be used to screen patients for common mental disorders and exclude patients with severe mental illness, substance use disorders, or suicidality. It will additionally be used to track metrics to determine Reach (i.e., number in need).

SECONDARY OUTCOMES:
Patient Health Questionnaire - 9 (PHQ-9) | measured at pre-treatment and weeks 8, 12, 20, 32
  The PHQ-9 is an instrument for screening, diagnosing, monitoring, and measuring severity of depression. Score cut offs for depression are 5 (mild), 10 (moderate), 15 (moderately severe) and 20 (severe).
Generalized Anxiety Disorder - 7 (GAD-7) | measured at pre-treatment and weeks 8, 12, 20, 32
  GAD-7 is a screening instrument with seven items to assess presence and severity of generalized anxiety severity. Scores range from 0 (not at all) to 3 (nearly every day) for a total range of 0 to 21. Score cut off points are 5 (mild), 10 (moderate), 15 (severe) anxiety.
PTSD Checklist - Civilian Version (PCL-C) | measured at pre-treatment and weeks 8, 12, 20, 32
  The PCL-C is a standardized self-report scale for PTSD comprised of 17 items. It uses a 5-point scale where respondents indicate how much they have been bothered by a symptom (1 = Not at All
  - 5 = Extremely). Items are totaled for a severity score (range = 17-85; 17-29 = little to no severity; 30-44 = moderate to moderately high severity; 45-85 = high severity).
Revised Conflict Tactics Scale | measured at pre-treatment and weeks 8, 12, 20, 32
  The Revised Conflict Tactics Scale measures physical, psychological, and sexual intimate partner violence. It consists of 39 items are asked twice: once for respondent and once for partner. Item responses gauge frequency and range from "Never" to "20 or more times." It has five subscales: Negotiation, Psychological Aggression, Physical Assault, Injury, and Sexual Coercion.
Dyadic Adjustment Scale | measured at pre-treatment and weeks 8, 12, 20, 32
  The Dyadic Adjustment Scale (32 Likert items) measures relationship functioning and satisfaction. The four subscales include: Dyadic Satisfaction, Dyadic Consensus, Dyadic Cohesion, and Dyadic Affectional Expression. The score range is 1-151. A higher score indicates better adjustment to marriage.
Alcohol Use Disorders Identification Test (AUDIT) | measured at pre-treatment and weeks 8, 12, 20, 32
  The AUDIT is comprised of 10 items that screen for hazardous or dependent drinking levels. Questions range from 0 to 4 with the exception of items 9 and 10 which have three response options and are scored 0, 2, 4. Items are summed. Score cut off points are 8 (hazardous drinking) and 13 women/15 men (alcohol dependence).

OTHER OUTCOMES:
Adverse Childhood Experiences-International Questionnaire | measured at pre-treatment
  The Adverse Childhood Experiences- International Questionnaire (43 dichotomous (yes/no) and Likert scale items) measures adverse childhood experiences. Domains include family dysfunction; physical, sexual and emotional abuse and neglect by parents or caregivers; peer violence; witnessing community violence; and exposure to collective violence. A higher composite score indicates more adverse experiences an individual was exposed to in childhood.